CLINICAL TRIAL: NCT00286663
Title: Evaluation of the Cellular Immune Response in Patients With Anti-SLA/LP- or Anti-LKM-Positive Autoimmune Hepatitis
Brief Title: Autoimmune Hepatitis Study
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator moving out of state, no other staff to lead research.
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Parvez S. Mantry, MD, University of Rochester Medical Center Liver and Digestive Disease Unit
Other Study IDs: RSRB 12494
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Last update posted 2008-07-09 (Estimated); Status verified 2008-07

CONDITIONS: Hepatitis, Autoimmune
Keywords: AIH, Autoimmune Hepatitis
MeSH Terms: conditions — Hepatitis, Autoimmune

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of the study is to determine the role special antibodies play in possibly identifying Autoimmune Hepatitis through the following:

Identify the response of specific T cells to antibodies and Monitor the response of the cells that regulate the immune system

DETAILED DESCRIPTION:
The object of this protocol is to characterize and monitor auto antigen-specific T cell responses in blood and liver biopsies of patients with anti-SLA/LP or anti-LKM-positive autoimmune hepatitis. The results will provide insight into the pathogenesis of autoimmune hepatitis and the monitoring of auto antigen-specific T cell reactivity in correlation to disease exacerbation and therapy.

ELIGIBILITY:
Inclusion Criteria:

Male or female subjects,All ethnic groups, Over 18 years of age, anti-SLA/LP or anti-LKM-positive autoimmune hepatitis

Exclusion Criteria:

Subjects with a hematocrit of <25

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-01; Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parvez S Mantry, MD, Principal Investigator — University of Rochester